CLINICAL TRIAL: NCT01411592
Title: Randomized Clinical Trial on Single Retainer All-Ceramic Resin-bonded Fixed Dental Protheses: Impact of the Bonding System
Brief Title: Single Retainer All-Ceramic Resin-bonded Fixed Dental Protheses
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Kiel (Other)
Collaborators: Ivoclar Vivadent AG (Industry)
Responsible Party: Principal Investigator, Martin Sasse, Dr. Martin Sasse, D.M.D., Assistant Professor, University of Kiel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ivoclar ZirCAD Adh.bruecken
Record Dates: First submitted 2011-08-03; First posted 2011-08-08 (Estimated); Results first posted 2014-09-11 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Restauration in Situ; Final Loss of Restauration; Debonded Restauration
Keywords: All-Ceramic; Resin-bonded Fixed Dental Protheses; Single Retainer; Randomized Clinical Trial; Resin Bond; Bonding System
MeSH Terms: interventions — multilink adhesive system; Metals

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Multilink (Active Comparator): RBFDPs were inserted using an adhesive bonding system with a phosphonic acid acrylate primer for the zirconia ceramic (Multilink-Automix bonding system [A/B primer and Multilink-Automix] with Metal/Zirconia primer)
  Interventions: Other: Multilink
- Panavia 21 TC (Active Comparator): RBFDPs were inserted using a phosphate monomer containing resin (Panavia 21 TC) without any primer
  Interventions: Other: Panavia 21 TC

INTERVENTIONS:
Other: Multilink — After air-abrasion of the retainer wings (50 µm alumina particles at 0.25 MPa) and etching the enamel with 36% phosphoric acid for 30 sec, the RBFDPs were inserted using an adhesive bonding system with a phosphonic acid acrylate primer for the zirconia ceramic (Multilink-Automix bonding system with Metal/Zirconia primer)
  Other Names: Multilink-Automix, Ivoclar Vivadent; Metal/Zirconia-Primer, Ivoclar Vivadent; A/B-Primer, Ivoclar Vivadent
  Arms: Multilink
Other: Panavia 21 TC — After air-abrasion of the retainer wings (50 µm alumina particles at 0.25 MPa) and etching the enamel with 36% phosphoric acid for 30 sec, the RBFDPs were inserted using a phosphate monomer containing resin (Panavia 21 TC) without any primer
  Other Names: Panavia 21 TC, Kuraray
  Arms: Panavia 21 TC

SUMMARY:
The purpose of this prospective study was to evaluate the clinical outcome of all-ceramic RBFDP with a cantilevered single-retainer design made from zirconia ceramic. To evaluate the impact of the adhesive system used an established resin cement with an integrated adhesive monomer (Panavia 21 TC) and a resin cement with a separate primer (Multilink Automix with Metal/Zirconia Primer) were compared within the study on a randomized basis.

The aim of the present randomized study was to evaluate wether the difference in bond strength of Panavia and Multilink Automix with Metal/Zirconia Primer to densely sintered zirconia ceramic (IPS e.max ZirCAD, Ivoclar Vivadent) has any impact on the clinical outcome of all-ceramic RBFDP with a cantilevered single-retainer design.

ELIGIBILITY:
Inclusion Criteria:

* sufficient oral hygiene
* one caries free or almost caries free abutment tooth available
* sufficient space for the retainer wing available
* patients willingness to return at regular intervals for at least 5 years for evaluation

Exclusion Criteria:

* clinical symptoms of bruxism
* collision, full or semi-contact sports (Boxing, Karate)
* pregnant women
* untreated advanced periodontitis

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-10; Primary Completion 2008-04 (Actual); Study Completion 2018-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Kern, DDS, PhD, Study Director — University of Kiel

REFERENCES:
- [Derived] Sasse M, Kern M. CAD/CAM single retainer zirconia-ceramic resin-bonded fixed dental prostheses: clinical outcome after 5 years. Int J Comput Dent. 2013;16(2):109-18. English, German. PMID 23930573

RESULTS

PARTICIPANT FLOW:
Groups:
- Multilink: 14 RBFDPs were inserted using an adhesive bonding system with a phosphonic acid acrylate primer for the zirconia ceramic (Multilink-Automix bonding system [A/B primer and Multilink-Automix] with Metal/Zirconia primer).
  Multilink bonding: After air-abrasion of the retainer wings (50 µm alumina particles at 0.25 MPa) and etching the enamel with 36% phosphoric acid for 30 sec, the RBFDPs were inserted using an adhesive bonding system with a phosphonic acid acrylate primer for the zirconia ceramic (Multilink-Automix bonding system with Metal/Zirconia primer).
  Patients were recalled after 6 and 12 months, and then annually.
- Panavia 21 TC: 16 RBFDPs were inserted using a phosphate monomer containing resin (Panavia 21 TC) without any primer.
  Panavia 21 TC: After air-abrasion of the retainer wings (50 µm alumina particles at 0.25 MPa) and etching the enamel with 36% phosphoric acid for 30 sec, the RBFDPs were inserted using a phosphate monomer containing resin (Panavia 21 TC) without any primer.
  Patients were recalled after 6 and 12 months, and then annually.
Period: Overall Study
Arm/Group | Multilink | Panavia 21 TC
Started | 14 | 16
5-Year Time Frame | 14 | 16
Completed | 14 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Multilink | Panavia 21 TC | Total
Number analyzed (Participants) | 14 | 16 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.57 (16.84) | 36.56 (20.36) | 33.3 (18.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 2 | 6 | 8
Region of Enrollment [Number; unit: participants]
  Germany | 14 | 16 | 30

OUTCOME MEASURES:

1. Primary Outcome: Final Loss of the Restauration
Time Frame: 5 years
Measure: Number; unit: participants
Arm/Group | Multilink | Panavia 21 TC
Number analyzed (Participants) | 14 | 16
participants | 0 | 0

2. Secondary Outcome: Debonding of the RBFDP
Description: Restoration was rebonded without any impairment of function
Time Frame: 5 years
Measure: Number; unit: participants
Arm/Group | Multilink | Panavia 21 TC
Number analyzed (Participants) | 14 | 16
participants | 1 | 1

ADVERSE EVENTS:
Arm/Group | Multilink | Panavia 21 TC
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/16
Other Adverse Events (participants affected / at risk) | 1/14 | 1/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Multilink (N=14) | Panavia 21 TC (N=16)
Debonding (Investigations) | 1 (1) | 1 (1) — Debonding of RBFDP. Treatment: Rebonding as initially conducted.
[Small Caries lesion] (Investigations) | 0 (0) | 1 (1) — Treatment: Composite resin filling.
[Rotation of abutment tooth] (Investigations) | 0 (0) | 1 (1) — Treatment: Derotated with a splint.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes